CLINICAL TRIAL: NCT06563700
Title: A Double Masked, Randomised, Longitudinal Comparative Study to Evaluate the Myopia Progression of Novel Spectacle Lenses Versus Single Vision Spectacle Lenses in Children With Myopia
Brief Title: Novel Lenses for Myopia Progression Trial
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Shanghai Eye Disease Prevention and Treatment Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2024-002
Record Dates: First submitted 2024-08-06; First posted 2024-08-21 (Actual); Last update posted 2025-12-03 (Actual); Status verified 2025-08

CONDITIONS: Myopia, Progressive
MeSH Terms: conditions — Myopia, Degenerative

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Group A (Placebo Comparator): single vision lens
  Interventions: Other: spectacle lens; Other: single vision lens
- Group B (Experimental): one of ZEISS BD spectacle lens designs 1 to 5
  Interventions: Other: spectacle lens
- Group C (Experimental): one of ZEISS BD spectacle lens designs 1 to 5
  Interventions: Other: spectacle lens
- Group D (Experimental): one of ZEISS BD spectacle lens designs 1 to 5
  Interventions: Other: spectacle lens
- Group E (Experimental): one of ZEISS BD spectacle lens designs 1 to 5
  Interventions: Other: spectacle lens
- Group F (Experimental): one of ZEISS BD spectacle lens designs 1 to 5
  Interventions: Other: spectacle lens

INTERVENTIONS:
Other: spectacle lens — one of ZEISS BD spectacle lens designs 1 to 5
Other: single vision lens — single vision lens
  Arms: Group A

SUMMARY:
This is a multi-center , prospective, randomised, longitudinal study to evaluate rate of myopia progression with novel lenses compared to Single-Vision spectacles. A total of 342 children will be recruited where 57 participants each are randomised to wear one of 5 test spectacle lens designs or a single vision lens (control) for 12 months. At the end of 12 months, those randomised to single vision lenses will be transferred to one of the test lenses and all the groups continued for another 12 months. Myopia progression during the second year with test lenses will be compared to historical or published controls.

ELIGIBILITY:
Inclusion Criteria:

be accompanied by a parent or guardian who is able to read and comprehend Chinese/English and sign a record of informed consent/assent; at baseline, be within the age range of 7 to 13 years old inclusive; be diagnosed as myopic having cycloplegic spherical equivalent between -0.75 dioptre (D) and -5.00 dioptre (D); astigmatism ≤1.50D; anisometropia of not more than 1.50D; be willing to comply with the wearing of clinical trial spectacles and clinical trial visit schedule as directed by the investigator; have ocular findings deemed to be normal; vision correctable to at least 0.8 or better in each eye with spectacles.

Exclusion Criteria:

Any pre-existing systemic or ocular condition, including infection or disease that is likely to affect visual acuity and refractive error; Any systemic disease that adversely affects ocular health e.g. diabetes, Graves disease, and auto-immune diseases such as ankylosing spondylitis, multiple sclerosis, Sjögrens syndrome and systemic lupus erythematosus. Conditions such as systemic hypertension and arthritis do not automatically exclude prospective participants.

Use of or a need for any systemic medication or topical medications which may alter normal ocular findings / are known to affect a participant's ocular health / physiology in an adverse or beneficial manner at enrolment and/or during the clinical trial.

History of eye trauma Amblyopia Strabismus History of use of myopia control interventions such as Orthokeratology, atropine or eye surgery 6 months prior to commencement of this trial.

Known allergy or intolerance to ingredients to cycloplegic eye-drops. Currently enrolled in another clinical trial.

Ages: 7 Years to 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 300 (Estimated)
Dates: Start 2024-08-16 (Actual); Primary Completion 2027-07-31 (Estimated); Study Completion 2027-07-31 (Estimated)

PRIMARY OUTCOMES:
myopia progression | 12 monthly
  change in spherical equivalent from baseline for each of the groups of BD test lenses and the single vision control group

SECONDARY OUTCOMES:
axial elongation | 12 monthly
  change in axial length from baseline for each of the groups of BD test lenses and the single vision control group
Subjective responses and compliance | 12 monthly
  Subjective visual responses of wearing spectacles and compliance using questionair for each groups

CONTACTS AND LOCATIONS:
Overall Officials: Xiangui He, Principal Investigator — Shanghai Eye Diseases Prevention and Treatment Center
Locations (1):
- Shanghai Eye Disease Prevention and Treatment Center, Shanghai, China